CLINICAL TRIAL: NCT00705627
Title: A Multicenter Trial Comparing Neoadjuvant Chemotherapy Followed by CCRT v.s. CCRT Alone in Locoregionally Advanced Nasopharyngeal Carcinoma
Brief Title: A Multicenter Trial Comparing Multi-course Chemotherapy in Locoregionally Advanced Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Guangdong Provincial People's Hospital (Other); Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other); Affiliated Cancer Hospital of Shantou University Medical College (Other)
Responsible Party: Principal Investigator, Hong Ming-huang, the director of GCP, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007047
Record Dates: First submitted 2008-06-24; First posted 2008-06-26 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-05

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: nasopharyngeal carcinoma; neoadjuvant chemotherapy; concurrent chemotherapy; randomized controlled clinical trials
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Neoadjuvant Therapy; Chemoradiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- B (Experimental): Drug: cisplatin. Patients in the control arm received radical radiotherapy, and cisplatin (80mg/m2 on day 1) every three weeks for three cycles during RT.
  Interventions: Drug: neoadjuvant chemotherapy plus concurrent chemoradiotherapy

INTERVENTIONS:
Drug: neoadjuvant chemotherapy plus concurrent chemoradiotherapy — Drug: cisplatin,fluorouracil. Patients received cisplatin 80mg/m2 on day 1,fluorouracil 4000mg/m2 civ 120 hours every three weeks for two cycles, then received radical radiotherapy, and cisplatin (80mg/m2 on day 1) every three weeks for three cycles during RT.
  Other Names: Neoadjuvant Chemotherapy Followed by CCRT

SUMMARY:
Locoregionally advanced nasopharyngeal carcinoma (NPC)(stage III, IV in UICC 2002 Classification) can be divided into two groups according to the risk of metastasis: high-risk metastasis group (T4 or N2-3) and low-risk metastasis group (T3N0-1). In low-risk metastasis group, concurrent chemoradiotherapy (CCRT) might decrease local recurrence and distance metastasis, which benefits overall survival. On the other hand, neoadjuvant chemotherapy is also associated with lower distance metastasis of advanced stage NPC. Nevertheless, CCRT alone or neoadjuvant chemotherapy alone leads to unsatisfactory results regarding to distance metastasis in patients with high-risk metastasis group. In this case, it is utmost important to investigate the new treatment combining neoadjuvant chemotherapy plus CCRT in order to improve overall survival of locoregionally advanced NPC with high-risk metastasis.

In our study, in order to investigate the effect and adverse reaction of neoadjuvant chemotherapy plus CCRT on distance metastasis and locoregionally relapse, four hundred patients with high risk of distance metastasis will be randomly divided into two groups, comparing neoadjuvant chemotherapy (DDP+5FU) plus CCRT (DDP) and CCRT (DDP) alone. We aim to find out the best therapeutic regimen with lowest adverse reaction for NPCS with high risk of distance metastasis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly histologically confirmed nasopharyngeal carcinoma, including WHO II or III
* Original clinical stage must be T4 or N2-3 （UICC 2002）
* Male and no pregnant female
* Age between 18-60
* WBC ≥4,000/mm3 and PLT ≥ 100,000/mm3
* With normal liver function test (ALT、AST≤2.5×ULN)
* With normal renal function test (Creatinine ≤ 1.5×ULN)
* Performance status scale ECOG grade 0，1
* Without radiotherapy or chemotherapy
* Patients must give signed informed consent

Exclusion Criteria:

* Patients have evidence of relapse or distant metastasis
* The presence of uncontrolled life-threatening illness
* Receiving other ways of anti-cancer therapy
* Receiving radiotherapy or chemotherapy
* Investigator consider the patients can't finish the whole study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2008-06; Primary Completion 2015-02 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
distant metastasis free survival,disease free survival | 5-Yr

SECONDARY OUTCOMES:
overall survival | 5-Yr

CONTACTS AND LOCATIONS:
Overall Officials: Minghuang Hong, MD, Study Chair — Sun Yet sen Cancer Center, China
Locations (1):
- Department of Nasopharyngeal Carcinoma, Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China